CLINICAL TRIAL: NCT03266419
Title: A Double-blind, Randomized, Parallel Design to Compare the Effectiveness of Deep Versus Moderate Neuromuscular Blockade With Standard-pressure Pneumoperitoneum During Laparoscopic Gastrectomy on Postoperative Pain in Surgical Patients
Brief Title: Effectiveness of Deep Versus Moderate Neuromuscular Blockade
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Byung-Moon Choi, Associate Profesor, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2017-0966
Record Dates: First submitted 2017-08-21; First posted 2017-08-30 (Actual); Results first posted 2019-11-13 (Actual); Last update posted 2019-11-13 (Actual); Status verified 2019-10

CONDITIONS: Neuromuscular Blockade

STUDY DESIGN:
Intervention Model Description: This study is investigator-initiated, randomized, double blinded clinical trial.
Who Masked: Participant, Outcomes Assessor
Masking Description: Researchers who evaluate postoperative pain will be blinded to the patient's allocation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Deep NMB using rocuronium (Experimental): The abdomen is insufflated to 13 mmHg pneumoperitoneum with deep NMB (post tetanic count 1-2) during operation
  Interventions: Drug: Deep NMB using rocuronium
- Moderate NMB using rocuronium (Active Comparator): The abdomen is insufflated to 13 mmHg pneumoperitoneum with moderate NMB (train of four 1-2) during operation
  Interventions: Drug: Moderate NMB using rocuronium

INTERVENTIONS:
Drug: Deep NMB using rocuronium — * Drug: rocuronium
  * Bolus dose: 0.7 mg/kg
  * Continuous infusion : 0.8-1.2 mg/kg/h for maintaining deep NMB (post tetanic count 1-2) during operation.
  Arms: Deep NMB using rocuronium
Drug: Moderate NMB using rocuronium — * Drug: rocuronium
  * Bolus dose: none
  * Continuous infusion: 0.2-0.6 mg/kg/h for maintaining moderate NMB (train of four 1-2) during operation.
  Arms: Moderate NMB using rocuronium

SUMMARY:
The aim of this study is to evaluate the influence of depth of neuromuscular blockade during laparoscopic gastrectomy on postoperative pain in surgical patients allocated randomly to either deep or moderate neuromuscular blockade group with standard-pressure pneumoperitoneum of 13 mmHg.

DETAILED DESCRIPTION:
* All patients were fasted from midnight without premedication
* Once in the operating room, the patients were monitored using electrocardiography, pulse oximetry, end-tidal carbon dioxide partial pressure, non-invasive blood pressure, and bispectral index (Aspect 2000; Aspect Medical Systems, Inc., Newton, MA, USA) measurements.
* Neuromuscular transmission was monitored using the M-NMT® module at the adductor pollicis muscle (Carescape® B850, GE Healthcare, Milwaukee, WI, USA).
* Throughout the surgery, these data were continuously downloaded to personal computers by using RS232C cables.
* Following pre-oxygenation with 100% O2, anesthesia was induced with propofol and remifentanil, which were administered using a target effect-site concentration-controlled infusion pump (Perfusor® Space, B. Braun Melsungen, Germany) by using the models suggested by Schnider et al. and Minto et al (Minto et al., 1997; Schnider et al., 1998).
* Tracheal intubation was facilitated with rocuronium 0.6 mg/kg.
* After tracheal intubation, the lungs of the patients were then ventilated with oxygen in air (1:1) and the ventilation rate was adjusted to maintain the end-tidal carbon dioxide partial pressure between 35 and 45 mmHg.
* For deep NMB group, an intravenous bolus of rocuronium (0.7 mg/kg) was given 2 minutes after intubation, followed by a continuous infusion of rocuronium of 0.8-1.2 mg/kg/h for maintaining deep NMB (post tetanic count 1-2) during operation. PTC was measured every 5 minutes. In the case of deviations from the target PTC, the pump speed could be increased or decreased or a bolus dose (10 mg) could be given.
* For moderate NMB group, no further loading dose of rocuronium was given. An intravenous infusion with rocuronium (0.2-0.6 mg/kg/h) was started at a TOF count of 1 for maintaining moderate NMB (train of four 1-2) during operation. TOF was measured every 5 minutes. In the case of deviations from the target TOF, the pump speed could be increased or decreased or a bolus dose (10 mg) could be given.
* The target effect-site concentrations of propofol were adjusted within a range of 2.5-3 μg/ml to maintain the bispectral index values at less than 60 during the induction and maintenance of anesthesia.
* The target effect-site concentrations of remifentanil were titrated to prevent signs of inadequate anesthesia and to maintain stable hemodynamics (SBP > 80 mmHg and HR > 45 beats/min).

  • Signs of inadequate anesthesia: systemic arterial blood pressure increased to greater than 15 mm Hg higher than the patient's normal value; heart rate exceeding 90 beats/min in the absence of hypovolemia; somatic responses, such as body movements (minimal muscle paralysis allowed physical movement), swallowing, coughing, grimacing, or opening of the eyes; and autonomic signs of inadequate anesthesia (Ausems, Vuyk, Hug, & Stanski, 1988)
* If necessary, ephedrine or atropine is administered to maintain systolic blood pressure above 80 mmHg and heart rate above 45 beats/min during anesthesia.
* An abdominal pressure of 13 mmHg was maintained during the laparoscopic surgery.
* When the surgeon asks for muscle relaxation due to the inability to obtain a visible laparoscopic field, additional bolus dose of rocuronium (10 mg) should be given.
* All patients were administered a bolus dose of oxycodone of 0.05 mg/kg at the end of pneumoperitoneum.
* IV PCA with oxycodone is started after the administration of loading dose. A semi-electronic pump (Automed 3200; Ace Medical, Seoul, South Korea) is used for PCA with demand bolus of 1 ml, background infusion of 1 ml/h and lock-out time of 15 min. The concentration of oxycodone in IV PCA bag is 1 mg/ml, and the volume of oxycodone-normal saline mixture delivered to patients for approximately 4 days is 200 ml.
* Rocuronium infusions are discontinued after deflation of CO2.
* After the end of surgery, a single intravenous bolus dose of sugammadex 2 or 4 mg/kg was administered for reversal of moderate and deep NMB, respectively.
* After the end of surgery, patients were taken to the PACU, and assessed for pain every 10 min using a VAS (0=no pain; 10=the most severe pain).
* Researchers who evaluate postoperative pain will be blinded to the patient's allocation
* Pain was measured at rest and when the wound areas were compressed with a force of 20 N (i.e., 2 kg of pressure imposed by three fingers on a 10 cm2 area). The wound compression was performed by a blinded researcher who was trained with an algometer (Commander Algometer, J Tech Medical Industries, Midvale, UT, USA) to apply this force consistently.
* The patient was administered intravenous oxycodone 2 mg (body weight <80 kg) or 3 mg (>80 kg) every 10 min until the VAS assessments showed that the pain intensity had decreased to <3 at rest and <5 on wound compression. At this point, MEAD of oxycodone was determined.
* VAS for wound and shoulder pain were also assessed at 6 and 24 h after the end of surgery.
* Postoperative nausea and vomiting were evaluated using the Rhodes index of nausea vomiting retching (RINVR) at 6 and 24 h after the end of surgery (Lee et al., 2016).
* After the end of surgery, the surgeon scored the surgical working conditions according to a five-point ordinal scale ranging from 1 (extremely poor conditions) to 5 (optimal conditions) (Martini et al., 2014).
* If the surgeon requests blind cessation for patient safety reasons, blindness is lifted.

ELIGIBILITY:
Inclusion Criteria:

* Patients 20 to 65 years old
* American Society of Anesthesiologist Physical Status 1, 2 or 3
* Patients undergoing laparoscopic gastrectomy
* Patients who signed a written informed consent form

Exclusion Criteria:

* Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive urine pregnancy test
* Patients with known hypersensitivity to rocuronium or sugammadex
* Patient with VAS score (0=no pain; 100=the most severe pain) of at least 10 before surgery
* Patients with liver cirrhosis confirmed by abdominal CT
* Patients with neuromuscular disease that may interfere with neuromuscular data (ex. Duchenne muscular dystrophy, myasthenia gravis)
* Clinically significant impairment of cardiovascular function, defined by ejection fraction < 50%
* Clinically significant impairment of renal function, defined by estimated GFR < 60 ml/min or need for hemodialysis
* Clinically significant impairment of liver function, defined by alanine aminotransferase > 100 IU/L
* Indication for rapid sequence induction
* Use of opioids within the 7 days prior to surgery
* History of abdominal surgery
* History of chronic obstructive pulmonary disease
* Body mass index (BMI) ≥ 35 kg/m2
* Body weight < 50 kg
* Conversion to laparotomy
* Family history of malignant hyperthermia
* Patients who are considered by the investigator to be unsuitable to participate in the study for any other reason not mentioned in the inclusion and exclusion criteria

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2018-03-28 (Actual); Primary Completion 2018-11-01 (Actual); Study Completion 2018-11-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Byung-Moon Choi, Dr, Principal Investigator — Department of Anesthesiology and Pain Medicine, Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No
Because MSD provides research funding, the IPD of this study will not be shared with other researchers.

REFERENCES:
- [Derived] Choi BM, Ki SH, Lee YH, Gong CS, Kim HS, Lee IS, Kim BS, Kim BS, Noh GJ. Effects of depth of neuromuscular block on postoperative pain during laparoscopic gastrectomy: A randomised controlled trial. Eur J Anaesthesiol. 2019 Nov;36(11):863-870. doi: 10.1097/EJA.0000000000001082. PMID 31503037

RESULTS

PARTICIPANT FLOW:
Groups:
- Deep NMB Using Rocuronium: The abdomen is insufflated to 13 mmHg pneumoperitoneum with deep NMB (post tetanic count 1-2) during operation
  Deep NMB using rocuronium: - Drug: rocuronium
  * Bolus dose: 0.7 mg/kg
  * Continuous infusion : 0.8-1.2 mg/kg/h for maintaining deep NMB (post tetanic count 1-2) during operation.
- Moderate NMB Using Rocuronium: The abdomen is insufflated to 13 mmHg pneumoperitoneum with moderate NMB (train of four 1-2) during operation
  Moderate NMB using rocuronium: - Drug: rocuronium
  * Bolus dose: none
  * Continuous infusion: 0.2-0.6 mg/kg/h for maintaining moderate NMB (train of four 1-2) during operation.
Period: Overall Study
Arm/Group | Deep NMB Using Rocuronium | Moderate NMB Using Rocuronium
Started | 51 | 49
Completed | 51 | 49
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Deep NMB Using Rocuronium | Moderate NMB Using Rocuronium | Total
Number analyzed (Participants) | 51 | 49 | 100
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 58 [49 to 63] | 58 [51 to 61] | 58 [51 to 62]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 16 | 32
  Male | 35 | 33 | 68
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  South Korea | 51 | 49 | 100
Duration of pneumoperitoneum [Median (Inter-Quartile Range); unit: minute] — Time taken to maintain pneumoperitoneum during operation (minute)
  minute | 117.0 [91.8 to 137.5] | 102.0 [88.0 to 120.5] | 109 [89 to 131.5]

OUTCOME MEASURES:

1. Primary Outcome: Minimum Effective Analgesic Dose (MEAD) of Oxycodone at Postoperative Care Unit (PACU)
Description: The patient was administered intravenous oxycodone 2 mg (body weight <80 kg) or 3 mg (>80 kg) every 10 min until the VAS (visual analogue scale)assessments showed that the pain intensity had decreased to <3 at rest and <5 on wound compression. At this point, MEAD of oxycodone was determined. The range of VAS is 0-10 (0 = no pain; 10 = most severe pain).
Time Frame: Through study period in PACU (post anesthesia care unit), up to 2 hours
Population: patients undergoing elective laparoscopic gastrectomy
Measure: Median (Full Range); unit: mg
Arm/Group | Deep NMB Using Rocuronium | Moderate NMB Using Rocuronium
Number analyzed (Participants) | 51 | 49
mg | 8.0 [2 to 26] | 8.0 [2 to 27]

2. Secondary Outcome: Mean Visual Analogue Scale (VAS) Score for Wound Pain at Post Anesthesia Care Unit (PACU)
Description: The patient was administered intravenous oxycodone 2 mg (body weight <80 kg) or 3 mg (>80 kg) every 10 min until the visual analogue scale (VAS) assessments showed that the pain intensity had decreased to <3 at rest and <5 on wound compression. At this point, the minimum effective analgesic dose (MEAD) of oxycodone was determined. The range of VAS is 0-10 (0 = no pain; 10 = most severe pain).
Time Frame: Through study period in post anesthesia care unit (PACU), an average of about 1 hour
Population: patients undergoing elective laparoscopic gastrectomy
Measure: Mean (Full Range); unit: mm
Arm/Group | Deep NMB Using Rocuronium | Moderate NMB Using Rocuronium
Number analyzed (Participants) | 51 | 49
mm | 6.1 [2.8 to 8.4] | 6.1 [2.7 to 7.3]

ADVERSE EVENTS:
Time Frame: postoperative 24 h
Arm/Group | Deep NMB Using Rocuronium | Moderate NMB Using Rocuronium
All-Cause Mortality (participants affected / at risk) | 0/51 | 0/49
Serious Adverse Events (participants affected / at risk) | 0/51 | 0/49
Other Adverse Events (participants affected / at risk) | 0/51 | 0/49

LIMITATIONS AND CAVEATS:
Pain assessment was performed only until 24 h after the end of surgery.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-18): https://cdn.clinicaltrials.gov/large-docs/19/NCT03266419/Prot_SAP_000.pdf